CLINICAL TRIAL: NCT06751264
Title: Evaluation of the Efficacy and Safety of Microwave Ablation of Uterine Adenomyosis Under Improved Ultrasound Guidance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Aerospace Center Hospital (Other)
Responsible Party: Principal Investigator, Liang Lei, Peking University Aerospace Centre Hospital, Peking University Aerospace Center Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-076
Record Dates: First submitted 2024-12-13; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Adenomyosis of Uterus
MeSH Terms: conditions — Adenomyosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Peritoneal water isolation (Experimental): Peritoneal water isolation
  Interventions: Procedure: Peritoneal water isolation
- Peritoneal combined with intrauterine water isolation (Experimental): Peritoneal combined with intrauterine water isolation
  Interventions: Procedure: Peritoneal combined with intrauterine water isolation

INTERVENTIONS:
Procedure: Peritoneal combined with intrauterine water isolation — On the basis of the conventional peritoneal water isolation group, the improved technology group added additional intrauterine water isolation, and continued to inject ice saline to separate the endometrium on both sides.
  Arms: Peritoneal combined with intrauterine water isolation
Procedure: Peritoneal water isolation — Transabdominal injection of saline into the abdominal cavity to achieve complete separation of the uterus from the surrounding organs and structures
  Arms: Peritoneal water isolation

SUMMARY:
This study aims to compare the safety and efficacy of segmental power adjustment combined with uterine cavity hydro-isolation in microwave ablation of adenomyosis

ELIGIBILITY:
Inclusion Criteria:

1. UFs or AM diagnosed by pathology and ultrasound；
2. Relevant symptoms such asabnormal uterine bleeding, secondary anemia, progressive dysmenorrhea and enlargement of the uterus；
3. Voluntarily undergo MWA；
4. a confirmed available safe transabdominal puncture path；

Exclusion Criteria:

1. Pregnancy or malignancy；
2. Severe and uncorrectable coagulation disorders；
3. Severe cardiac, liver, and renal dysfunction；
4. Anesthesia allergy.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — female
Enrollment: 137 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The rates of endometrial injury | From enrollment to the end of treatment at 3 months
  Observe the differences in the rates of endometrial injury between two groups

SECONDARY OUTCOMES:
The reduction rate of adenomyosis volume | From enrollment to the end of treatment at 1 year
  Observe the reduction rate of adenomyosis volume between two groups
complication | From enrollment to the end of treatment at 1 year
  The complication rate between the two groups was compared

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: ICF, CSR